CLINICAL TRIAL: NCT00360828
Title: A Phase II Study of Irinotecan HCI in Patients With Recurrent Anaplastic Astrocytomas, Mixed Malignant Gliomas, and Oligodendrogliomas
Brief Title: Phase II Study of Irinotecan HCI for Recurrent Anaplastic Astrocytomas, Mixed Malignant Gliomas, and Oligodendrogliomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator left Moffitt and study had low accrual.
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MCC-14633
Record Dates: First submitted 2006-08-03; First posted 2006-08-07 (Estimated); Results first posted 2011-12-09 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2011-11

CONDITIONS: Astrocytoma; Glioma; Oligodendroglioma
Keywords: Recurrent Anaplastic Astrocytoma; Mixed Malignant Glioma; Oligodendroglioma; Irinotecan; Brain tumor; Nitrosoureas; Brain and nervous system
MeSH Terms: conditions — Astrocytoma; Glioma; Oligodendroglioma; Brain Neoplasms; Neurologic Manifestations | interventions — Irinotecan; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irinotecan Treatment (Experimental): Participants were given irinotecan at a fixed dose: [350 mg/m2 in patients either not on anti-seizure drugs or on anti-seizure drugs which do not interfere with the metabolism of Irinotecan; 600 mg/m2 in patients on anti-seizure drugs which interfere with the metabolism of Irinotecan] once every 21 days. Depending on how many side effects were experienced with the first cycle [first 21 days], the dose of both drugs may remain the same or may be decreased to make the treatment better tolerated with less side effects. The irinotecan was given to through a vein over 90 minutes.
  Interventions: Drug: Irinotecan Hydrochloride (HCI) Treatment; Drug: Continued Irinotecan Hydrochloride (HCI) Treatment

INTERVENTIONS:
Drug: Irinotecan Hydrochloride (HCI) Treatment — Irinotecan injections. Irinotecan hydrochloride [CPT-11; CAMPTOSAR] is an antineoplastic agent of the topoisomerase I inhibitor class. The drug is supplied in amber vials and appears as a pale yellow transparent aqueous solution. Two vial sizes are available: 2 mL vials containing 40 mg of drug and 5 mL vials containing 100 mg of drug. A treatment cycle was 21 days. Patients were treated for a minimum of 3 cycles (doses) of CPT-11 or until their disease progressed.
  Other Names: CPT-11; CAMPTOSAR; Irinotecan HCL
Drug: Continued Irinotecan Hydrochloride (HCI) Treatment — For patients responding to treatment, therapy could have continued beyond 18 cycles.
  Other Names: CPT-11; CAMPTOSAR; Irinotecan HCL

SUMMARY:
Phase 2 trial to explore the efficacy and safety of irinotecan (CPT-11). Also administered at each cycle was zofran/Kytril/Anzemet, decadron, and IV atropine.

At each cycle, patient exams and interviews as well as lab results were to help the research team to determine the symptomatic side effects of the treatment. Recorded past toxicities were to be compared with current side effects.

DETAILED DESCRIPTION:
Phase 2 trial to explore the efficacy and safety of irinotecan (CPT-11) in patients with recurrent anaplastic astrocytomas (AA), mixed malignant glioma, and oligodendrogliomas (OA). Patients were to be stratified by tumor histology and treated with CPT-11 every 21 days (treatment cycle).

Baseline data (collected <14 days) was to consist of a neurological/oncological history, neurological examination, height, weight, performance status, Quality Of Life FACT-L questionnaire, laboratory studies to include complete blood count (CBC), differential, platelets, prothrombin time (PT), complete metabolic panel (CMP), Lactose dehydrogenase (LDH), and a pregnancy test, as well as a cranial Computerized Tomography/Magnetic Resonance Imaging (CT/MRI) with and without contrast (to measure or evaluate the size and location of the tumor before treatment).

Administered every 21 days was a dose of irinotecan (CPT-11), zofran/Kytril/Anzemet, decadron, and intravenous (IV) atropine. At each cycle, patient exams and interviews as well as lab results were to help the research team to determine the symptomatic side effects of the treatment. Recorded past toxicities were to be compared with current side effects.

Between days 15-21 (within 7 days of next scheduled CPT-11 treatment) the following tests were to be repeated - a neurological/oncological history and neurological examination, weight, blood drawn (CMP, LDH), performance status, and Quality Of Life FACT-L questionnaire. Also, a MRI (Cranial CT/MRI with and without contrast) was to be performed for tumor assessments at week 9, 18, 27, 36, and after every nine weeks thereafter until progression. Response was to be measured by a reduction in tumor size.

These supportive therapies were provided as necessary:

* Antiemetic Therapy
* Anticholinergics
* Loperamide (Imodium®)
* Growth Factors
* Other Concomitant Medications

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological or neuroradiographic documented recurrent glioma defined as an anaplastic astrocytoma, mixed malignant glioma or oligodendroglioma. All patients must have had prior pathologic confirmation of primary tumor histology.
* Patients must be > than or equal to 18 years old.
* Patients must have a Karnofsky performance score (KPS) of > or equal to 50
* Measurable disease per MacDonald criteria is required
* Patients must have a predicted life expectancy of at least 12 weeks
* Required initial laboratory data:

  1. Absolute Neutrophil Count (ANC) > 1,500
  2. Platelets > 100,000
  3. Serum Creatinine < 2.0
  4. Serum Bilirubin < 2.0
  5. Aspartamine transaminase/ Alanine transaminase (AST/ALT) < 3x normal
  6. Pregnancy test for females with child-bearing potential negative
* Patients must sign and date an IRB approved informed consent form stating he or she is aware of the neoplastic nature of the disease. Patient must willingly provide written consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts. (Human protection committee approval of this protocol and consent form is required).
* Patients must be willing and able to comply with scheduled visits, treatment plan, and laboratory tests and accessible for follow-up.
* Patients must have been previously treated with both surgery and radiotherapy.
* Prior adjuvant and one salvage chemotherapy regimen is permitted.
* Prior stereotactic radiotherapy is permitted.

Exclusion Criteria:

* Patients have evidence of leptomeningeal spread of disease.
* Patients having been treated with 2 or more salvage regimens.
* Pregnant or breast-feeding women. With the exception of post-menopausal or infertile women, a negative blood test for pregnancy is mandatory before entry on study. Fertile persons refusing to use adequate contraceptives may not participate.
* Patients with a history of irritable bowel disease, irritable bowel syndrome, chronic diarrhea or presence of a bowel obstruction.
* Patients with a second active malignancy or diagnosis of other cancer within 3 years of enrollment, except for surgically cured basal cell carcinoma, or in situ carcinoma of the cervix.
* Mentally incapacitated patients or psychiatric illness that would prevent the patient from giving informed consent.
* Patients with poorly controlled diabetes, hepatitis infection, uncontrolled high blood pressure, unstable angina, symptomatic congestive heart failure, and myocardial infarction within the previous six months, or serious uncontrolled cardiac arrhythmia.
* Known to be human immunodeficiency virus (HIV) positive or to have an acquired immunodeficiency syndrome (AIDS) related illness.
* Patients with an active infection that is not adequately controlled with antibiotics.
* Patients with other severe concurrent disease, which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Patients with a known sensitivity to any of the products to be administered during treatment.
* Patients currently enrolled in another clinical trial or patients who have participated in a trial of an investigational device or drug within the last 30 days.
* Patients previously treated with CPT-11.
* Concurrent stereotactic radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Pan, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://www.moffitt.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 12 consented, 2 were not eligible after the screening process.
Groups:
- Irinotecan Hydrochloride (HCI) Treatment: Participants were given irinotecan at a fixed dose: [350 mg/m2 in patients either not on anti-seizure drugs or on anti-seizure drugs which do not interfere with the metabolism of Irinotecan; 600 mg/m2 in patients on anti-seizure drugs which interfere with the metabolism of Irinotecan] once every 21 days. Depending on how many side effects were experienced with the first cycle [first 21 days], the dose of both drugs may remain the same or may be decreased to make the treatment better tolerated with less side effects. The irinotecan was given to through a vein over 90 minutes.
Period: Overall Study
Arm/Group | Irinotecan Hydrochloride (HCI) Treatment
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Irinotecan Hydrochloride (HCI) Treatment
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response After 3 Cycles of Treatment
Description: The intent was to have 63 evaluable participants to determine the Objective Response Rate utilizing Criteria for Response, Progression and Relapse according to the McDonald Criteria. A measurement is made of the maximal enhancing tumor diameter on a single axial gadolinium-enhanced T1-weighted section, and then the largest perpendicular diameter is measured on the same image. The product of the 2 diameters is calculated, and the measurements are repeated with each scan. Measurements from multiple lesions are summed.
Time Frame: 3 cycles (21 day cycles)
Population: All participants having stable disease
Measure: Number; unit: participants
Arm/Group | Irinotecan Hydrochloride (HCI) Treatment
Number analyzed (Participants) | 10
participants | 8

2. Secondary Outcome: Overall Survival at 6 Months
Description: Patients surviving 6 months after treatment end
Time Frame: 6 months post treatment end
Population: All participants who received at least one dose of drug
Measure: Number; unit: participants
Arm/Group | Irinotecan Hydrochloride (HCI) Treatment
Number analyzed (Participants) | 10
participants | 6

3. Secondary Outcome: Progression Free Survival
Description: Patients surviving at one year post treatment end
Time Frame: 1 year post treatment end
Population: The low accrual rate prevented us from completing the planned analysis.
Arm/Group | Irinotecan Hydrochloride (HCI) Treatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Frequency and Severity of Toxicity
Description: Toxicities assessed through 3 months
Time Frame: 3 months
Population: The low accrual rate prevented us from completing the planned analysis.
Arm/Group | Irinotecan Hydrochloride (HCI) Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival at 12 Months
Description: Patients surviving 12 months after last dose of drug
Time Frame: 12 months post treatment end
Population: All participants who received at least one dose of drug
Measure: Number; unit: participants
Arm/Group | Irinotecan Hydrochloride (HCI) Treatment
Number analyzed (Participants) | 10
participants | 6

ADVERSE EVENTS:
Time Frame: 1 year, 9 months
Arm/Group | Irinotecan Hydrochloride (HCI) Treatment
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irinotecan Hydrochloride (HCI) Treatment (N=10)
Diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 3, definitely related.

LIMITATIONS AND CAVEATS:
Low accrual prevented us from completing the planned analysis. The initial Principal Investigator (PI) left Moffitt and there were only 10 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No